CLINICAL TRIAL: NCT06830655
Title: Functional and Performance Determinants in Climbers: Examining the Role of Mobility, Stability, and Fatigue Across Proficiency Levels
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Principal Investigator, Bartosz Wilczyński, Scientists, PhD, Medical University of Gdansk
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: NKB/530/2024
Record Dates: First submitted 2025-01-31; First posted 2025-02-17 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Fatigue; Joint Hypermobility Syndrome; Climbing Injuries; Cognitive Fatigue
Keywords: Bouldering; Sports Performance Assessment; Climbing-Specific Performance; Hand Grip Strength; Indoor Climbing; Outdoor Climbing
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will not be informed about the study's hypotheses comparing elite and intermediate climbers or the specific effects of fatigue on their performance. This ensures that participants perform to the best of their abilities without bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Professional Climbers (Experimental): Pre- and post-intervention assessment of the fatigue protocol.
  Interventions: Other: Fatigue Protocol
- Amateur Climbers (Experimental): Pre- and post-intervention assessment of the fatigue protocol.
  Interventions: Other: Fatigue Protocol
- Indoor Climbers (Experimental): Pre- and post-intervention assessment of the fatigue protocol.
  Interventions: Other: Fatigue Protocol
- Outdoor Climbers (Experimental): Pre- and post-intervention assessment of the fatigue protocol.
  Interventions: Other: Fatigue Protocol

INTERVENTIONS:
Other: Fatigue Protocol — After the warm-up, each participant will be assigned the easiest route of their skill level on the "Kilter Board" with a 15-degree wall incline. Participants will start the route from the initial holds and finish it with the need to touch the top hold with both hands. They will be instructed to climb as quickly and smoothly as possible. After reaching the last hold, they will descend along the same route to the initial holds without touching the ground. The procedure will be repeated until the participant reports fatigue that prevents further climbing. Any stoppage by the participant during the protocol will not be allowed to last longer than 5 seconds, will be recorded, and categorized as either isometric contraction or rest time, depending on the nature of the stoppage, which will be established during records analyzing.

SUMMARY:
The primary objective is to understand how motor skills and fatigue affect climbing performance in indoor and outdoor climbers, also comparing elite and amateur climbers.

Aims:

* Assess differences in selected joint range of motion, isometric strength, and dynamic stability between elite and intermediate climbers.
* Evaluate the impact of the fatigue protocol on functional performance and cognitive outcomes across climbers of varying skill levels (intermediate vs. advanced).
* Examine the impact of general joint hypermobility, as indicated by Beighton Scores, on functional climbing performance.
* Association between cognitive factors (e.g., attention, memory) and motor skills.

Research questions:

* Do elite climbers have better joint mobility and balance than amateur climbers?
* How does fatigue affect performance and reaction time and cognitive function?
* Does having flexible joints (joint hypermobility) make climbers better athletes
* What are the performance differences between indoor and outdoor climbers?

This study will help identify key skills and physical traits that improve climbing performance. It will also explore how fatigue and flexibility impact safety and performance in different climbing environments.

DETAILED DESCRIPTION:
Detailed Description

This study investigates the functional and performance determinants in indoor and outdoor climbers, focusing on mobility, stability, fatigue, and skill level. The protocol will compare elite and intermediate climbers through various physical and cognitive assessments conducted before and after a climbing-specific fatigue protocol. The goal is to identify key biomechanical, physiological, and cognitive factors that influence climbing performance and fatigue resistance in both climbing environments.

ELIGIBILITY:
Inclusion Criteria:

* primary sport discipline - climbing (bouldering/lead rock or other)
* Healthy (without injury, pain, or symptoms) at the time of the study
* Participation in climbing training (minimum 3 months)

Exclusion Criteria:

* pain or other symptoms related during study
* rheumatological disease
* neurological disease or balance disorders
* orthopaedic disease
* genetic disease
* cardiovascular system disease
* surgeries of upper and lower limb in the last year
* surgeries of spine in the last year
* a primary sport other than climbing.
* taking medications that may affect balance.
* use of orthopedic supplies during the study

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Dynamic Balance (Y-Balance Test) Lower and Upper Quarter | through study completion, an average of 2 years
  The test will be performed for both the lower and upper body. For the lower body, the participant will begin by standing with one foot on the center foot plate. While maintaining a single-leg stance, the participant will reach with the free leg in one of three directions (anterior, posteromedial, and posterolateral) three times, then repeat the process with the opposite leg. The procedure will then be repeated for the remaining directions. The maximal reach distance in each direction will be measured and included in the analysis. For the upper body, the participant will begin by up position of a push up. While maintaining a single-arm push up, the participant will reach with the free arm in on of three directions (medial, inferolateral and superolateral) "cm". Test will be assesed before and after fatigue protocol.
ISOMETRIC STRENGTH TEST - Shoulder Internal and External Rotation | through study completion, an average of 2 years
  Isometric strength assessments of shoulder internal and external rotations will be conducted using the Lafayette Hand-Held Dynamometer (HHD). Participants will be positioned appropriately, in prone and then supine with the shoulder abducted to 90 degrees. The dynamometer will be placed just proximal to the wrist. Participants will be instructed to exert maximal force against the device for a specified duration, 5 seconds. This process will be repeated for multiple trials to ensure consistent and reliable measurements. The Lafayette HHD will provide objective data on muscle strength, facilitating the evaluation and monitoring of participant progress throughout the study. Results will be expressed in newtons (N) or normalized to body weight as newtons per kilogram (N/kg).
ISOMETRIC STRENGTH TEST - Pinching | through study completion, an average of 2 years
  Pinching a dynamometer. The participant will be seated with the elbow fully extended and the shoulder positioned at 0° flexion. The task will involve exerting maximum force, with separate trials performed for the dominant and non-dominant hand. The dynamometer will be held between the thumb and fingers to measure the force generated, with results recorded in units of force. The emphasis will be on achieving maximum effort to ensure reliable and consistent results. In "kg"

SECONDARY OUTCOMES:
RANGE OF MOTION (Shoulder Internal and External Rotation) | through study completion, an average of 2 years
  The participant will lie in a supine position with the shoulder positioned at 90° of abduction and aligned with the plane of the glenoid. Researcher 1 will palpate the coracoid process while passively moving the humerus into internal rotation. Researcher will apply the HALO digital goniometer ((Halo, Halo Medical Devices, Subiaco, Western Australia) to the proximal part of the forearm. The measurement will be taken at the point when movement of the coracoid process is first detected, indicating the limit of passive glenohumeral internal rotation and the onset of scapular motion. The angle of rotation will be measured in degrees.Shoulder External Rotation: The participant will lie in a supine position with the shoulder positioned at 90° of abduction and aligned with the plane of the glenoid.
RANGE OF MOTION (Passive Ankle dorsiflexion range of motion (Gastrocnemius muscle flexibility test) | through study completion, an average of 2 years
  The participant will lie in a supine position with the knee straight and the ankle joint positioned off the table. Researcher 1 will test the maximum dorsiflexion of the foot while controlling the position of the knee. Researcher 2 will apply the HALO digital goniometer (Halo, Halo Medical Devices, Subiaco, Western Australia) to the outer edge of the foot. The angle of dorsiflexion will be measured in degrees.
Active Ankle Dorsiflexion range of motion (The Weight Bearing Lunge Test (WBLT)) | through study completion, an average of 2 years
  Participants were positioned facing a wall, with the test foot placed at a predetermined distance. The knee was advanced toward the wall until it lightly contacted the surface, ensuring the heel remained in contact with the ground. The distance between the big toe and the wall was adjusted to determine the participant's maximum dorsiflexion range, which was subsequently recorded as the measured distance from the big toe to the wall (cm).
Hypermobility - Beighton score | through study completion, an average of 2 years
  The test consisted of the abduction of the thumb to the forearm, the knee hyperextension above 10 degrees, the extension of the metacarpophalangeal joint in the 5th finger above 90 degrees, the elbow hyperextension above 10 degrees, and the placing flat hands on the floor. Each positive test scored 1 point.
Climbing specific foot rise | through study completion, an average of 2 years
  The participant will stand on both footholds with feet placed hip-width apart, and hands gripping the rung at shoulder-width apart. The rung will be set at the participant's head height, rounded to the nearest 5 cm. The participant will raise one foot as high as possible along the scale, with the leg either straight or slightly flexed at the knee. The test will be performed in two variations: with rotation, where natural rotation of the shoulders and hips is allowed, and without rotation, where the shoulders and hips must remain parallel to the wall. The height of the foot rise will be measured in centimeters.
Hand-eye response time test | through study completion, an average of 2 years
  A-Champs ROX Pro (A-Champs Interactive Training Solutions, S.L., Spain) system will be used to measure hand-eye response time. Each participant will perform the test three times with both their dominant and non-dominant hand with the best time recorded as the participant's response time in milliseconds. Four discs will be positioned on the floor and arranged in a square formation, spaced 1.5 meters apart. Participants will lie in a prone position at a distance that allows them to comfortably reach all discs based on their arm length. Participants will be instructed to deactivate each illuminated disc as quickly as possible by tapping it with the hand being tested. The test will run for 30 seconds, with discs lighting up in a random order and will automatically end after the 30-second test period.
Power slap | through study completion, an average of 2 years
  The participant will hang from a designated rung with arms fully extended above the head, knees bent and feet positioned behind the body. The participant will use open finger grip, with the thumb permitted to rest on the rung. The task will involve performing an explosive pull-up without momentum, releasing the dominant hand to slap as high as possible. The result of the test, measured as the height of the slap, will be recorded in centimeters.
Finger hang test | through study completion, an average of 2 years
  The participant will grip a designated rung with arms fully extended and shoulders aligned to their natural width. Feet must remain off the ground throughout the test. The participant will use open finger grip, with the thumb permitted to rest on the rung. The researcher will closely monitor the participant's grip, ensuring proper starting and hanging posture. Endurance time will be recorded in seconds using a stopwatch, starting from the initiation of the hang and stopping when grip failure occurs. To maintain consistency across participants, only one trial will be conducted per individual.

OTHER OUTCOMES:
Participants characteristics - Body Mass Index | through study completion, an average of 2 years
  weight and height will be combined to report BMI in kg/m^2
Cognitive Tests - Corsi-block task (total score, %) | through study completion, an average of 2 years
  Corsi-block task (PEBL; Mueller & Piper). Visuospatial working memory test. During the retrieval period, participants were instructed to immediately reproduce the same sequence of blue squares in the same order as they were presented. Corsi Span - The maximum number of blocks correctly recalled in the correct order before failure (reported as a whole number, e.g., 4). Accuracy (%) - The percentage of correctly recalled sequences.
Cognitive Tests - Corsi-block task - Reaction Time (RT, in milliseconds) | through study completion, an average of 2 years
  Corsi-block task (PEBL; Mueller & Piper). Visuospatial working memory test. During the retrieval period, participants were instructed to immediately reproduce the same sequence of blue squares in the same order as they were presented. Reaction Time (RT, in milliseconds) - Time taken to begin recalling the sequence.
Cognitive Tests - STROOP - (Accuracy (%)) | through study completion, an average of 2 years
  STROOP. Cognitive control and selective attention, measuring the ability to manage cognitive interference. Participants will be presented with color words (e.g., "red," "blue") displayed in various ink colors. They will be instructed to name the ink color, disregarding the word's meaning. This task will measure their ability to manage cognitive interference. Accuracy (%) - Percentage of correct responses.
Cognitive Tests - STROOP - Reaction Time (RT, in milliseconds, ms) | through study completion, an average of 2 years
  STROOP. Cognitive control and selective attention, measuring the ability to manage cognitive interference. Participants will be presented with color words (e.g., "red," "blue") displayed in various ink colors. They will be instructed to name the ink color, disregarding the word's meaning. This task will measure their ability to manage cognitive interference. Reaction Time (RT, in milliseconds, ms) - Time taken to correctly name the ink color.
Participants characteristics - Sports experience | through study completion, an average of 2 years
  Sports experience (years, months)
Participants characteristics - Sport workload (hours per trainings or competition) | through study completion, an average of 2 years
  Sports and training volume (hours per trainings or competition, weekly)
Participants characteristics - History of sports-related injuries | through study completion, an average of 2 years
  Questionaire - Question about sports-related injuries within sports career (sports participating in trainings and competitions) which included:
  * exact type of injury (acute or chronic, contact or non-contact)
  * location of injury (anatomic site, e.g. knee)
  * duration of injury (time-loss, in days)

CONTACTS AND LOCATIONS:
Overall Officials: Bartosz Wilczyński, PhD, Principal Investigator — Medical University of Gdansk; Mateusz Nowosad, Principal Investigator — Medical University of Gdansk
Locations (2):
- Poland (2):
  - Department of Immunobiology and Environment Microbiology, Medical University of Gdańsk, Gdansk, Gdańsk
  - Department of Immunobiology and Environment Microbiology, Medical University of Gdańsk, Gdansk

IPD SHARING:
Plan to Share IPD: No